CLINICAL TRIAL: NCT04937270
Title: Effects of High-frequency Deep Diathermy on Heart Rate Variability in Women With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, Researcher, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-1040781-A-N-012021046HR
Record Dates: First submitted 2021-06-09; First posted 2021-06-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Primary Dysmenorrhea; Dysmucorrhea

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High frequency application time is 5 minutes (Experimental): The group which treats for 5 minutes by using the high-frequency therapy device
  Interventions: Device: High frequency therapy (5 minutes)
- High frequency application time is 7 minutes (Experimental): The group which treats for 7 minutes by using the high-frequency therapy device
  Interventions: Device: High frequency therapy (7 minutes)
- High frequency application time is 9 minutes (Experimental): The group which treats for 9 minutes by using the high-frequency therapy device
  Interventions: Device: High frequency therapy (9 minutes)
- Superficial heat therapy (Active Comparator): Group treated with superficial heat therapy for 20 minutes
  Interventions: Device: Superficial heat therapy

INTERVENTIONS:
Device: High frequency therapy (5 minutes) — The high-frequency therapy device (radio frequency therapy, WINBACK, Villeneuve Loubet France) used in this study was used to treat deep heat for 5 minutes using a 500 kHz resistive electric transfer (RET).
  Arms: High frequency application time is 5 minutes
Device: High frequency therapy (7 minutes) — The high-frequency therapy device (radio frequency therapy, WINBACK, Villeneuve Loubet France) used in this study was used to treat deep heat for 7 minutes using a 500 kHz resistive electric transfer (RET).
  Arms: High frequency application time is 7 minutes
Device: High frequency therapy (9 minutes) — The high-frequency therapy device (radio frequency therapy, WINBACK, Villeneuve Loubet France) used in this study was used to treat deep heat for 9 minutes using a 500 kHz resistive electric transfer (RET).
  Arms: High frequency application time is 9 minutes
Device: Superficial heat therapy — In the physical therapy used in this study, it was applied for 20 minutes using conventionally used superficial heat therapy.
  Arms: Superficial heat therapy

SUMMARY:
Superficial heat therapy is mainly used to relieve menstrual pain, but it does not penetrate deeper than the skin tissue. In order to penetrate deep into the deep layers and promote tissue relaxation, deep heat therapy can be effective. The treatment time for deep heat treatment is controversial, and there is no study on deep heat treatment using radio frequency for dysmenorrhea. Therefore, in this study, by applying radiofrequency waves at different times to the lower abdomen for patients with primary dysmenorrhea, the pain and changes in the autonomic nervous system were compared with thermotherapy to suggest appropriate therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-50
* Regular menstrual cycle (24-32 days)
* Those who have had symptoms of primary dysmenorrhea for at least 1 year
* Those who have lower back pain symptoms related to menstrual pain of 5 or higher on the Visual Analysis Scale (VAS)
* The body mass index is between 20-30

Exclusion Criteria:

* pelvic inflammatory disease
* uterine fibroids, polycystic ovary syndrome. Those with gynecological findings such as endometriosis
* Those who have used an intrauterine contraceptive device
* Those who took birth control pills or nonsteroidal anti-inflammatory drugs at the time of the experiment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | immediate change after intervention in baseline
  Autonomic nervous system balance tester (SA3000new, Medicore Co. Korea) was used. The subjects placed electrodes on three areas (left arm, left leg, right leg) while lying down and performed for 3 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- The wells neuropain clinic, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes